CLINICAL TRIAL: NCT00689182
Title: A Phase II Trial of the Safety and Efficacy of Iron Reduction by Phlebotomy in Recipients of Hematopoietic Stem Cell Transplants
Brief Title: Safety and Efficacy of Iron Reduction by Phlebotomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea Kew (Other)
Responsible Party: Sponsor-Investigator, Andrea Kew, Dr., Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA017
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Iron Overload
Keywords: iron reduction; iron overload; phlebotomy; hematopoietic stem cell transplant
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All patients will receive phlebotomy
  Interventions: Procedure: monthly phlebotomy x 12 months

INTERVENTIONS:
Procedure: monthly phlebotomy x 12 months — All patients will receive monthly phlebotomies.

SUMMARY:
Hypothesis: The reduction of total body iron by phlebotomy will be safe and feasible in the post-HSCT setting

Iron overload is common after hematopoietic stem cell transplantation. It is associated with chronic liver disease, with increased rates of infection and decreased survival.

Eligible, consenting patients will have once monthly phlebotomy procedures (500ml) for 12 months.

SAFETY: At each visit, patients will have a comprehensive assessment prior to starting and after completing the phlebotomy. This assessment will include determination of pain at phlebotomy site, local infection and an assessment of symptoms of anemia including presyncope, fatigue and dyspnea. The patient's pulse, blood pressure, respiratory rate and temperature will also be determined before and following the phlebotomy.

EFFICACY: Iron stores will be measured serially in each patient. Measurements will be performed prior to the start of phlebotomy, and at 6 months and 12 months following the start of the series of 12 phlebotomies. These evaluations will be undertaken regardless of the number of phlebotomies which the patient actually undergoes. Iron stores will be estimated by measuring serum ferritin and transferrin saturation levels. Total body iron will be estimated from hepatic and cardiac iron concentration as measured by magnetic resonance imaging (MRI). Gandon et al. (12) described a non-invasive technique using MRI to measure hepatic iron stores. Iron is a paramagnetic substance which causes local magnetic field inhomogeneities leading to dephasing and signal loss in MRI. Gradient echo sequences are most susceptible to their effects because they do not use a 180° refocusing pulse, unlike conventional spin-echo sequences. Gandon et al. used multiple gradient echo sequences, compared the signal in liver to adjacent muscle and used this ratio to correlate with hepatic iron levels measured on tissue biopsy samples using spectrophotometric analysis. Multiple sequences were used because the nomogram comparing the L/M signal ratio is linear over only a small concentration of tissue iron.

DETAILED DESCRIPTION:
Background Hematopoietic stem cell transplantation (HSCT) is increasingly used as a treatment for a variety of malignant and non-malignant conditions. With improvements in conditioning regimens and post-transplant care, more HSCT recipients are becoming long-term survivors and therefore increasing attention is being directed to studying the long-term consequences of successful HSCT.

Iron overload is surprisingly common after HSCT. The pathophysiology of iron overload or siderosis is related to transfusional iron, inhibition of normal erythropoiesis and released iron stores from hepatocytes, tumour cells and bone marrow. It is associated with chronic liver disease in this patient population, as well as with increased rates of infection. Studies suggest that iron overload may also affect survival in this population, as has been shown in other populations who are susceptible to iron overload such as those with thalassemia and hereditary hemochromatosis (1,2).

McKay et al. described 76 survivors of allogeneic and autologous HSCT who were at least 1 year post-transplant (3). Sixty-seven (88%) had a ferritin level above the normal range. Thirty-one (41%) had abnormal liver enzymes and 30/31 also had elevated ferritin. At the time of publication, 10 of the patients had begun a venesection program; all showed a reduction in ferritin levels and nine patients had a reduction in alanine aminotransferase (ALT). Strasser et al. showed an increase of hepatic iron concentration in 10 consecutive patients who died post-HSCT (4). In a retrospective study to determine the characteristics of chronic liver disease post-HSCT, iron overload was felt to contribute to chronic liver dysfunction in 52.4% of patients post-HSCT who had liver disease (5).

Iron overload has also been associated with an increased frequency of infection in HSCT recipients. A single-centre retrospective study of autopsies conducted post-HSCT revealed an association between high liver iron concentration and invasive Aspergillus infection (6). In a consecutive series of 263 allogeneic HSCT patients, 5 cases of mucormycosis all occurred in patients with severe iron overload (7).

Iron overload prior to transplantation may also have a negative effect on survival. In a prospective study of 25 consecutive patients, Altes et al. showed that a very high ferritin level and a high transferrin saturation prior to conditioning was associated with a decreased overall survival and a high transferrin saturation was associated with an increase in transplant-related mortality (8).

Therapeutic phlebotomy is well-established for treatment of iron overload associated with hereditary hemochromatosis (9) and beta thalassemia after HSCT (10). Phlebotomy has also been studied in survivors of acute leukemia with iron overload. Franchini et al. showed that phlebotomy was feasible and well-tolerated in this population and resulted in normalization of ferritin and transferrin saturation (11). This study demonstrated feasibility of phlebotomy but the effect of iron reduction on end-organ function was not addressed.

In summary, iron overload is common following HSCT and has been associated with a number of adverse biochemical and clinical outcomes. In other clinical settings such as hereditary hemochromatosis and transfusional iron overload states such as thalassemia, the reduction of iron stores by phlebotomy or chelation has been unequivocally demonstrated to reduce both morbidity and mortality. We therefore postulate that the reduction of iron overload after HSCT will similarly be associated with lower morbidity and mortality.

Objectives

1. demonstrate the safety and feasibility of phlebotomy to reduce total body iron in HSCT recipients
2. demonstrate reduction in total body iron by reduced ferritin and transferrin saturation and reduction in hepatic and cardiac iron
3. demonstrate improvements in end-organ function by improved hepatic, cardiac and endocrine function.

Study Design This is a prospective, single arm phase II trial designed to evaluate the safety and efficacy of decreasing total body iron in HSCT recipients by phlebotomy.

Study Intervention Patients who are eligible to participate and who give informed consent will undergo a regimen of phlebotomy in the following manner. Starting after 60 days post-transplant, the patients will undergo a phlebotomy of 500 mL of whole blood monthly for a total of 12 treatments. There will be a determination of the complete blood count prior to each phlebotomy and if the hemoglobin level is less than 100 g/L, the phlebotomy will not be performed. Patients will not routinely receive crystalloid volume replacement following the phlebotomy. However, if a patient experiences syncope or pre-syncope, subsequent phlebotomies will be followed by the infusion of 500 mL of normal saline.

Assessment of Safety and Feasibility The safety and feasibility of regular phlebotomy will be determined by assessing the proportion of patients who can complete the 12 planned phlebotomies. Delays in phlebotomy and reasons for stopping the phlebotomy program will be documented. At each visit, patients will have a comprehensive assessment prior to starting and after completing the phlebotomy. This assessment will include determination of pain at phlebotomy site, local infection and an assessment of symptoms of anemia including presyncope, fatigue and dyspnea. The patient's pulse, blood pressure, respiratory rate and temperature will also be determined before and following the phlebotomy.

Assessment of Adverse Events and Serious Adverse Events In this study, only those adverse events felt to be related to study procedures will be recorded. Phlebotomy adverse events include: Pain at phlebotomy site, infection at phlebotomy site, evidence of phlebitis, fatigue, presyncope, syncope, dyspnea, bacteremia, cellulitis at the phlebotomy site. A fall in systolic blood pressure of greater than 20 mmHg post-phlebotomy will also be considered an adverse event.

Only serious adverse events related to study procedures will be recorded.

Patients will be carefully assessed before and after the phlebotomy procedure. Adverse events and serious adverse events related to study procedures will be assessed throughout the study and up to 30 days following the last phlebotomy.

Assessment of Efficacy Determination of iron concentration Iron stores will be measured serially in each patient. Measurements will be performed prior to the start of phlebotomy, and at 6 months and 12 months following the start of the series of 12 phlebotomies. These evaluations will be undertaken regardless of the number of phlebotomies which the patient actually undergoes. Iron stores will be estimated by measuring serum ferritin and transferrin saturation levels. Total body iron will be estimated from hepatic and cardiac iron concentration as measured by magnetic resonance imaging (MRI). Gandon et al. (12) described a non-invasive technique using MRI to measure hepatic iron stores. Iron is a paramagnetic substance which causes local magnetic field inhomogeneities leading to dephasing and signal loss in MRI. Gradient echo sequences are most susceptible to their effects because they do not use a 180° refocusing pulse, unlike conventional spin-echo sequences. Gandon et al. used multiple gradient echo sequences, compared the signal in liver to adjacent muscle and used this ratio to correlate with hepatic iron levels measured on tissue biopsy samples using spectrophotometric analysis. Multiple sequences were used because the nomogram comparing the L/M signal ratio is linear over only a small concentration of tissue iron.

The accuracy of the MRI technique was subsequently verified by Alustiza et al. (13). They measured hepatic iron concentration in 112 patients with iron levels that varied from normal (n=68) to abnormal in patients with hereditary hemochromatosis (n=21) and transfusional hemosiderosis (n=23). The correlation coefficient between iron measured by MRI compared to tissue biopsy in this series was 0.957. This positive correlation verifies the Gandon technique.

Serum samples will also be collected at baseline to screen for the most common mutations of the HFE gene (C282Y mutation and H63D mutation) as hereditary hemochromatosis is common in the general population and may contribute to iron overload in HSCT recipients. The patient and family physician will be informed about the results of hemochromatosis testing and standard practice will be followed.

Determination of end organ function The effect of iron overload will be studied in three principal areas: liver, heart and endocrine organs. All measurements will be performed at baseline and at 6 and 12 months following the start of the series of 12 phlebotomies. Hepatic function will be determined by measurement of liver enzymes (alkaline phosphatase, aspartate aminotransferase and alanine aminotransferase) and liver function testing including total bilirubin, albumin and INR. Cardiac function will be determined by magnetic resonance imaging and serum brain natriuretic peptide and troponin. Endocrine function will be determined by measurement of serum LH, FSH, TSH, free T4, testosterone (males) and fasting glucose.

Follow-up After completion of the trial, patients will continue to be followed by their hematologist. If the phlebotomy is safe and feasible, their physician may choose to continue with phlebotomy but this would not be standard practice and there is not evidence to support the intervention at this time.

Analysis The analysis of the results of this study will be descriptive. A screening log will be kept and the number of patients screened for this study will be recorded. Patients who are eligible to participate and who give informed consent will be described according to the following parameters: age, gender, underlying indication for transplant, type of transplant, number of red cell transfusions received prior to transplant, number of red cell transfusions from the start of conditioning until study enrollment and ECOG performance status at time of study entry. The feasibility of the intervention will be recorded by describing the proportion of patients who complete the planned series of 12 phlebotomies. In order to consider the patients who are unable to complete all 12 phlebotomies, the total number of actual phlebotomies conducted in the trial will also be recorded and expressed as a proportion of the total number of planned phlebotomies. The number of phlebotomies per patient per time period will also be reported. The efficacy of the intervention will be recorded by describing the changes in serum ferritin and transferrin saturation, liver enzymes and liver function, endocrine parameters and liver and cardiac iron stores as determined by liver MRI. Cardiac function will also be determined at study entry and 6 and 12 months following the start of the series of 12 planned phlebotomies. The safety of the intervention will be recorded by evaluating the number of patients who had adverse and/or serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients who have undergone autologous or allogeneic HSCT
* who are red-cell transfusion-independent
* at least 60 days post-transplant
* serum ferritin of at least 1000ug/L
* ECOG less than or equal to 2.0

Exclusion Criteria:

* pregnancy
* breast-feeding
* serious infection
* HIV antibody positive
* renal failure (creatinine < 30ml/min)
* sever obstructive lung disease
* have a pacemaker, cerebral aneurysm or metal prosthesis
* evidence of disease relapse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Iron stores, total body iron | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kew, MD, Principal Investigator — Queen Elizabeth II Health Sciences Centre
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided